CLINICAL TRIAL: NCT00121901
Title: Does Glyceryl Nitrate Prevent Post-Endoscopic Retrograde Cholangiopancreaticography (ERCP) Pancreatitis?
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EPEPPS-06-2005
Record Dates: First submitted 2005-06-30; First posted 2005-07-21 (Estimated); Last update posted 2007-10-18 (Estimated); Status verified 2007-10

CONDITIONS: Pancreatitis
Keywords: Pancreatitis; Cholangiopancreatograpy, Endoscopic Retrograde/adverse; Nitroglycerin; Randomized Controlled Trial,
MeSH Terms: conditions — Pancreatitis

INTERVENTIONS:
Drug: glyceryl nitrate

SUMMARY:
Post-ERCP pancreatitis can be a serious complication to ERCP. Two studies have shown a promising preventive effect of glyceryl nitrate. This study should provide a final answer to the clinical question: Does glyceryl nitrate prevent post-ERCP pancreatitis? The study is a prospective, randomized, double blind, placebo-controlled multicenter trial. The investigators intend to include 1600 patients from Norway, Sweden, Denmark, and France.

The patients will receive either placebo or a glyceryl nitrate patch (15 mg/24 hours). Follow-up will occur after 7 days. The primary outcome measure will be post-ERCP pancreatitis, and secondary outcome measures will be mild, moderate and severe pancreatitis; post procedure pancreatitis-related mortality; and adverse events.

DETAILED DESCRIPTION:
Project:

This study will compare glyceryl nitrate (GN) treatment to non-active treatment for the prevention of post-ERCP acute pancreatitis, which is an inflammation of the pancreas that can occur after a procedure known as ERCP.

Background:

ERCP (endoscopic retrograde cholangiopancreaticography) is an examination of the pancreas by which it is possible to perform therapeutic measures such as stone removal from the common bile duct and visualisation of the pancreas. Inflammation of the pancreas after the ERCP procedure (called: post-ERCP pancreatitis) is the most feared and common complication of the ERCP. It occurs in 1-40% of patients, with rates of 5% or more being more typical. Currently, the background of post-ERCP pancreatitis is poorly known.

Attempts at preventing post-ERCP pancreatitis have been carried out through a change to low-risk techniques, by avoiding high-risk patients, and by use of pharmacological prophylaxis.

Glyceryl Nitrate:

Glyceryl nitrate is a well-known medicine used for many years in other diseases. Possible side effects are headache and low blood pressure. Other side effects such as dizziness, tiredness, nausea, local redness at the application site and allergic reactions of the skin are rare.

Aim:

The purpose of this study is to document that pre-treatment with GN is effective in preventing post-ERCP pancreatitis. In two earlier GN studies, sample sizes were relatively small (less than one hundred) and the rates of post-ERCP pancreatitis in the control group were quite high (15-17%). Therefore, further studies are needed to confirm the promising effect of GN in the prophylaxis of post-ERCP pancreatitis.

Participants:

The study includes every patient undergoing ERCP above the age of 18 years. Patients are excluded if they have active acute pancreatitis, previous sphincterotomy (cut in the sphincter at the end of the biliary and pancreatic ducts in the duodenum) or chronic pancreatitis with calcifications. Also, patients may not take sildenafil (Viagra) as GN should not be taken together with sildenafil. Patients allergic to glyceryl nitrate or glue should not be included. Patients with constrictive pericarditis (inflammation and fibrosis in the sack around the heart); pericardial tamponade (blood or liquor in the sack around the heart); low blood pressure; aortic stenosis (stenosis of the aortic valve); hypertrophic obstructive cardiomyopathy (a special disease with thickness of the heart); mitral stenosis (stenosis of the mitral valve); anemia (low hemoglobin); and untreated hypothyroidism (thyroid disease) are excluded because these are other diseases to which glyceryl nitrate should not be used. Pregnant women are excluded. Patients can only be included once.

Practical:

Patients have been preparing for the study as if it was a normal procedure. Prior to the procedure, patients will be asked to participate in the study. If the patients accept, after oral and written consent, they will receive either a GN patch or non-active patch on the chestwall 40-60 minutes prior to the ERCP procedure.

A canula is inserted in a cubital vein for medication. The ERCP is initiated, and patients are observed afterwards according to local practice, which is typically 3 hours. Patients are asked to fill out a letter with questions related to symptoms of pancreatitis (pain, fever, nausea, vomiting, hospitalization) to send to the investigating center after 7 days. If patients do not send the letter they will be contacted by phone within 14 days.

Interim analysis:

An interim analysis will be made, when 800 patients have been included. The study will stop, if 1) the interim analysis shows a significant higher mortality in one group than in the other or 2) if the study has proceeded more than 2 years.

Economy:

The project is a multicenter trial of the European Post-ERCP Pancreatitis Preventing Study Group. This local project is located at XX-department. No commercial interests are involved. The investigators/authors work for free against authorship. Finances are sought through funds for research.

References:

1. Freeman M. Post-ERCP pancreatitis: patient and technique-related risk factors. JOP 2002;3(6):169-176.
2. Demols A, Deviere J. New frontiers in the pharmacological prevention of post-ERCP pancreatitis: the cytokines. JOP 2003; 4(1):49-57.
3. Testoni P. Preventing post-ERCP pancreatitis: where are we?. JOP 2003; 4(1):22-32.
4. Mariani A. Pharmacological prevention of post-ERCP pancreatitis:which therapy is best?. JOP 2003; 4(1):68-74.
5. Murray B, Carter R et al. Diclofenac reduces the incidence of acute pancreatitis after endoscopic retrograde cholangiopancreatography. Gastroenterology 2003; 124:1786-1791.
6. Sand J, Nordback I. Prospective randomized trial of the effect of nifedipine on pancreatic irritation after endoscopic retrograde cholangiopancreatography. Digestion 1993; 54:105-11.
7. Sudhindran S, Bromwich E et al. Prospective randomized double-blind placebo-controlled trial of glyceryl trinitrate in endoscopic retrograde cholangiopancreaticography-induced pancreatitis. British J of Surg 2001; 88:1178-1182.
8. Moreto M, Zaballa M. et al. Transdermal glyceryl trinitrate for prevention of post-ERCP pancreatitis: a randomized double-blind trial. Gastrointest Endoscopy 2003;57:1-7.
9. Harrison et al. Bioequivalence comparison of two drug-in-adhesive transdermal nitroglycerine patches. Am J Ther 1996;3:580-585.
10. Pande H, Thuluvath PJ. Pharmacological prevention of post-endoscopic retrograde cholangiopancreatography pancreatitis. Drugs 2003;63(17):1799-1812.
11. Freeman ML. Prevention of post-ERCP pancreatitis: Pharmacologic solution or patient selection and pancreatic stents? Gastroenterology 2003;124(7):1977-1980.
12. Cotton PB, Lehman G, Vennes J, Geenen JE, et al. Endoscopic sphincterotomy complications and their management: an attempt at consensus. Gastrointest Endosc 1991;37:383-393.

ELIGIBILITY:
Inclusion Criteria:

* All patients (men and women) more than 18 years old who are going to have an ERCP procedure performed at the different centers from September 1, 2004 to about January 31, 2005 will be included.

Exclusion Criteria:

* Before the study: active acute pancreatitis (defined as: acute upper abdominal pain and S-amylases x 3 upper normal limit OR upper abdominal pain + radiological findings [CAT-/MR-scan] consistent with acute pancreatitis OR pathoanatomical findings consistent with acute pancreatitis by surgery)
* Known previous sphincterotomy
* Chronic pancreatitis with known calcifications
* Hypotension (definition: systolic blood pressure < 100 mmHg)
* Anemia, men/women (hemoglobin < 6 mmol/l or <9.7 g/dl)
* Constrictive pericarditis
* Pericardial tamponade
* Hypertrophic obstructive cardiomyopathy, aortic stenosis
* Mitral stenosis sildenafil within 24 hours before the ERCP procedure and 24 hours after the procedure
* Hypersensibility to nitroglycerine
* Hypersensibility to the applied glue on the patch
* Known untreated hypothyroidism
* Pregnancy or a potential to become pregnant, i.e. those who are not using safe contraception (intrauterine device [IUD] or oral contraception)
* Included earlier in the study
* Exchange of stent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2004-10; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
acute pancreatitis within 7 days after the ERCP procedure. (An independent committee at each center will retrospectively judge whether patients have had post-ERCP pancreatitis or not in respect to a specific definition.)

SECONDARY OUTCOMES:
mild, moderate, and severe pancreatitis as a criterion proposed by Cotton et al [12]
post procedure pancreatitis-related mortality
adverse events (severe and non-severe such as headache, dizziness, hypotension, hypersensibility, and others)

CONTACTS AND LOCATIONS:
Overall Officials: Camilla Nøjgaard Nøjgaard, MD, Principal Investigator — Gastroenheden, Hvidovre Hospital, Kettegård Alle 30, 2650 Hvidovre
Locations (14):
- Denmark (6):
  - Department of Medical and Surgical Gastroenterology, KAS Glostrup, Copenhagen, Glostrup
  - Dept. of Medical Gastroenterology F, KAS Gentofte, Copenhagen, Hellerup
  - Gastroenheden, Hvidovre Hospital, Copenhagen, Hvidovre
  - Rigshospitalet, Copenhagen, København Ø
  - Køge County Hospital, Køge, Køge
  - Dept of Medical Gastroenterology S, Odense Universitetshospital, Odense, Odense
- France (2):
  - Serv Gastroenterologie Hopital Sainte Marguerite, Marseille, Marseille Cedex 09
  - North Hospital, Marseille, Marseille
- Norway (4):
  - Div of Gastroenterology, dept. of Int Medicine Affiliated Hospital University of Oslo, Østfold Fredrikstad, Fredrikstad, Fredrikstad
  - Helse Fonna HF Haugesund Sjukehus Kirurgisk - vest blokk gastro, Haugesund, Haugesund
  - Ullevål Hospital, Oslo, Oslo County
  - Stavanger Hospital, Stavanger, Stavanger
- Sweden (2):
  - Halmstad Hospital, Halmstad, Halmstad
  - Dept of Surgery, University Hospital Malmö, Malmo, Malmö

REFERENCES:
- [Result] Freeman ML. Post-ERCP pancreatitis: patient and technique-related risk factors. JOP. 2002 Nov;3(6):169-76. No abstract available. PMID 12432183
- [Result] Demols A, Deviere J. New frontiers in the pharmacological prevention of post-ERCP pancreatitis: the cytokines. JOP. 2003 Jan;4(1):49-57. PMID 12555016
- [Result] Testoni PA. Preventing post-ERCP pancreatitis: where are we? JOP. 2003 Jan;4(1):22-32. PMID 12555013
- [Result] Mariani A. Pharmacological prevention of post-ERCP pancreatitis: which therapy is best? JOP. 2003 Jan;4(1):68-74. PMID 12555018
- [Result] Murray B, Carter R, Imrie C, Evans S, O'Suilleabhain C. Diclofenac reduces the incidence of acute pancreatitis after endoscopic retrograde cholangiopancreatography. Gastroenterology. 2003 Jun;124(7):1786-91. doi: 10.1016/s0016-5085(03)00384-6. PMID 12806612
- [Result] Sand J, Nordback I. Prospective randomized trial of the effect of nifedipine on pancreatic irritation after endoscopic retrograde cholangiopancreatography. Digestion. 1993;54(2):105-11. doi: 10.1159/000201021. PMID 8319838
- [Result] Sudhindran S, Bromwich E, Edwards PR. Prospective randomized double-blind placebo-controlled trial of glyceryl trinitrate in endoscopic retrograde cholangiopancreatography-induced pancreatitis. Br J Surg. 2001 Sep;88(9):1178-82. doi: 10.1046/j.0007-1323.2001.01842.x. PMID 11531863
- [Result] Moreto M, Zaballa M, Casado I, Merino O, Rueda M, Ramirez K, Urcelay R, Baranda A. Transdermal glyceryl trinitrate for prevention of post-ERCP pancreatitis: A randomized double-blind trial. Gastrointest Endosc. 2003 Jan;57(1):1-7. doi: 10.1067/mge.2003.29. PMID 12518122
- [Result] Harrison LI, Riedel DJ, Machacek JH, Crowley JK, Kanniainen CM, Hoglin JA, Robison TS, Zumhofe JM. Bioequivalence Comparison of Two Drug-in-Adhesive Transdermal Nitroglycerin Patches. Am J Ther. 1996 Aug;3(8):580-585. doi: 10.1097/00045391-199608000-00006. PMID 11862294
- [Result] Pande H, Thuluvath P. Pharmacological prevention of post-endoscopic retrograde cholangiopancreatography pancreatitis. Drugs. 2003;63(17):1799-812. doi: 10.2165/00003495-200363170-00003. PMID 12921486
- [Result] Freeman ML. Prevention of post-ERCP pancreatitis: pharmacologic solution or patient selection and pancreatic stents? Gastroenterology. 2003 Jun;124(7):1977-80. doi: 10.1016/s0016-5085(03)00553-5. No abstract available. PMID 12806633
- [Result] Cotton PB, Lehman G, Vennes J, Geenen JE, Russell RC, Meyers WC, Liguory C, Nickl N. Endoscopic sphincterotomy complications and their management: an attempt at consensus. Gastrointest Endosc. 1991 May-Jun;37(3):383-93. doi: 10.1016/s0016-5107(91)70740-2. PMID 2070995
- [Derived] Nojgaard C, Hornum M, Elkjaer M, Hjalmarsson C, Heyries L, Hauge T, Bakkevold K, Andersen PK, Matzen P; European Post-ERCP Pancreatitis Preventing Study Group. Does glyceryl nitrate prevent post-ERCP pancreatitis? A prospective, randomized, double-blind, placebo-controlled multicenter trial. Gastrointest Endosc. 2009 May;69(6):e31-7. doi: 10.1016/j.gie.2008.11.042. PMID 19410035